CLINICAL TRIAL: NCT03147729
Title: Radiofrequency in Anal Incontinence: Randomized Clinical Trials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, Juliana Barros Ferreira, Physical therapist, Escola Bahiana de Medicina e Saude Publica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 43462915.8.0000.554 4
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Radiation Exposure
Keywords: Radiofrequency; Anal incontinence; Fecal incontinence; Women sexual function; Sexuality
MeSH Terms: conditions — Encopresis; Fecal Incontinence; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiofrequency in anal incontinence: a pilot study (Other): It will be a single arm study with a group of anal incontinence with 10 women with anal incontinence
  Interventions: Radiation: Radiofrequency non ablation

INTERVENTIONS:
Radiation: Radiofrequency non ablation — Use of radiofrequency

SUMMARY:
Anal incontinence (AI) is used to englobe the involuntary loss of both fecal material and gases, which can help to improve quality of life. Based on these experiences objectives were drawn: to evaluate the effectiveness of radiofrequency and it's influence on quality of life of patients with anal incontinence, to correlate the anal incontinence severity and to evaluate a sexual function and to verify an influence with radiofrequency treatment. It is a blind randomized clinical trial. For the collection of data it was used a fecal quality of life questionnaire (FIQL). The questionnaire assess the severity of Anal Incontinence (FISI), the degree of patient's satisfaction using a five-point scale (Likert) and a visual analogue EVA scale). It was divided in two groups, in one group it was used radiofrequency and pelvic exercises and in the other turned off radiofrequency (heated glycerin) and pelvic exercises. It was accomplished in eight sections. As a result, it is expected the efficiency of the treatment of radiofrequency in the quality of life, in sexual function and in it's severity.

ELIGIBILITY:
Inclusion Criteria:

- Individuals between 18 and 66 years of age with a clinical complaint of Anal Incontinence and who agree to participate voluntarily in the research.

Exclusion Criteria:

* Individuals with cognitive impairment, use of pacemakers, women who use the Intra-Uterine Device (IUD) of copper, pregnant women, individuals who are taking vasodilators or anticoagulants and hemophiliacs, patients with cognitive deficits or psychiatric illness, patients with chronic neurological degenerative diseases and individuals with hemorrhoid metallic clamp.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of radiofrequency in anal incontinence | 8 radiofrequency sessions will be performed, with a 7 day interval between them. The session will be 20 minutes.Participants will be followed up for a minimum of 12 months.
  The radiofrequency application protocol will be used in the form of a capacitive electric transfer, bipolar configuration, with the Tonderm brand, Spectra G2 model, which has two electrodes: one active, in the anal region, with liquid glycerin and another, dispersive, coupled to the patient's hip. The temperature will be measured through a digital thermometer with infra-red until it reaches 41°C and will be maintained for 2 minutes. It will use Consent form, questionnaire of socio-demographic data and basic anamnesis. Then Fecal Incontinence Quality of Life, Fecal Incontinence Severity Index and Female Sexual Function Index. After, a perineal physical evaluation will be performed by an experienced Physical Therapist. The professional will perform a perineal muscle strength test, reflex and sensitivity test. For the sensitivity evaluation will be used a digital osiometer. The patients will be divided into two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola bahiana de Medicina e Saúde Pública, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Publication in scientific articles.